CLINICAL TRIAL: NCT00088634
Title: A Double-blind Fixed-dose Study of Lurasidone (SM-13496) and Placebo in the Treatment of Schizophrenia
Brief Title: A Study to Test the Effectiveness and Safety of a New Medication in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1050196
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lurasidone (Experimental): 80 mg AM dosing once daily
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone — 80 mg AM dosing once daily
  Arms: Lurasidone
Drug: Placebo — Matching Placebo to 40mg lurasidone tablets
  Arms: Placebo

SUMMARY:
A 6-week in-patient and out-patient study to test the effectiveness and safety of a new medication in the treatment of schizophrenia

DETAILED DESCRIPTION:
Study will evaluate the efficacy of a new compound versus placebo in the treatment of patients with schizophrenia (diagnosed by DSM-IV criteria) as measured by reductions from baseline on the total score of the Brief Psychiatric Rating Scale (BPRS) as extracted from the Positive and Negative Syndrome Scale (PANSS).

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV criteria for schizophrenia as established by SCID-CV
* The patient must agree to a voluntary hospitalization duration of 31 days minimum at the start of the treatment
* If female, must not be pregnant, or must be incapable of conceiving or be taking steps to prevent conception

Exclusion Criteria:

* The patient has used an investigational drug within the past 30 days
* The patient has participated in a previous study of this compound

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2004-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (22):
- United States (22):
  - Birmingham Psychiatry Pharmaceutical, Birmingham, Alabama
  - Summit Research Group, Little Rock, Arkansas
  - Comprehensive NeuroScience, Cerritos, California
  - Collaborative Neuro Science Network, Inc., Garden Grove, California
  - Optimum Health Services, La Mesa, California
  - California Clinical Trials, San Diego, California
  - CNRI, LLC San Diego, San Diego, California
  - Pacific Clinical Research, Upland, California
  - Comprehensive NeuroScience, Inc, Washington D.C., District of Columbia
  - Segal Institute for Clinical Research, North Miami, Florida
  - The Segal Institute, North Miami, Florida
  - University of South Florida, Department of Psychiatry and Behavioral Medicine, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive Neuroscience, Inc., Hoffman Estates, Illinois
  - Robert Lynn Horne, MD, Suite 4, Las Vegas, Nevada
  - CNS Research Institute, Clementon, New Jersey
  - Quantum Clinical Services Group, Philadelphia, Pennsylvania
  - Community Clinical Research, Austin, Texas
  - Future Search Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - InSite Clinical Research, DeSoto, Texas
  - CBH Health, L.L.C - Dominion Hospital, Falls Church, Virginia

REFERENCES:
- [Result] Nakamura M, Ogasa M, Guarino J, Phillips D, Severs J, Cucchiaro J, Loebel A. Lurasidone in the treatment of acute schizophrenia: a double-blind, placebo-controlled trial. J Clin Psychiatry. 2009 Jun;70(6):829-36. doi: 10.4088/JCP.08m04905. Epub 2009 Jun 2. PMID 19497249
- [Derived] Hopkins SC, Tomioka S, Ogirala A, Loebel A, Koblan KS, Marder SR. Assessment of Negative Symptoms in Clinical Trials of Acute Schizophrenia: Test of a Novel Enrichment Strategy. Schizophr Bull Open. 2022 Apr 7;3(1):sgac027. doi: 10.1093/schizbullopen/sgac027. eCollection 2022 Jan. PMID 39144777
- [Derived] Hopkins SC, Ogirala A, Worden M, Koblan KS. Depicting Safety Profile of TAAR1 Agonist Ulotaront Relative to Reactions Anticipated for a Dopamine D2-Based Pharmacological Class in FAERS. Clin Drug Investig. 2021 Dec;41(12):1067-1073. doi: 10.1007/s40261-021-01094-7. Epub 2021 Nov 9. PMID 34751928
- [Derived] Nasrallah HA, Cucchiaro JB, Mao Y, Pikalov AA, Loebel AD. Lurasidone for the treatment of depressive symptoms in schizophrenia: analysis of 4 pooled, 6-week, placebo-controlled studies. CNS Spectr. 2015 Apr;20(2):140-7. doi: 10.1017/S1092852914000285. Epub 2014 Jun 23. PMID 24955752

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 80 mg: 2 40 mg lurasidone tablets taken once/day
- Placebo: Matching placebo to lurasidone 40 mg tablets taken once/day
Period: Overall Study
Arm/Group | Lurasidone 80 mg | Placebo
Started | 90 | 90
Completed | 52 | 47
Not Completed | 38 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 80 mg | Placebo | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (9.91) | 41.9 (9.78) | 40.8 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 68 | 70 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Double-blind Treatment in the BPRS (Brief Psychiatric Rating Scale) Total Score
Description: The BPRS consists of 18 ordered categorical items (from "not present" to "extremely severe," on a 1- to 7-point scale), each developed to assess patient symptomatology in a relatively discrete symptom area. The BPRS will be extracted from the PANSS by adding the scores of the 18 items (P2 to P7, N1, N2, and G1 to G10) of the PANSS and will not be assessed separately.
Time Frame: Baseline and 6 weeks
Population: Efficacy analyses will be based on the ITT (intent-to-treat)population. The ITT population will consist of all patients who are randomized, taken one dose of study medication and had at least 1 post-baseline efficacy assessment of the PANSS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 90 | 90
units on a scale | -8.9 [-11.5 to -6.2] | -4.2 [-6.9 to -1.5]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Placebo; Comparisons between SM-13496 and placebo will be performed by means of a 2-way analysis of covariance (ANCOVA) model with treatment group and study center as factors, and baseline BPRS score as a covariate. Ninety-five percent (95%) confidence intervals will be constructed using the variability estimates from the ANCOVA model; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the PANSS (Positive and Negative Syndrome Scale) Scores
Description: The PANSS is a 30-item scale that evaluates positive, negative, and other symptoms in patients with schizophrenia. Each item is rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme). Scores range from 30-210 with higher scores representing a worsening of schizophrenia.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 90 | 90
units on a scale | -14.1 [-18.3 to -9.9] | -5.5 [-9.8 to -1.2]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Placebo; Comparisons between SM-13496 and placebo will be performed by means of a 2-way analysis of covariance (ANCOVA) model with treatment group and study center as factors, and baseline PANSS score as a covariate. Ninety-five percent (95%) confidence intervals will be constructed using the variability estimates from the ANCOVA model; Test type: Superiority or Other; p < 0.05, ANCOVA

3. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the CGI-S (Clinical Global Impression of Severity) Scores
Description: The CGI Severity (CGI-S) assesses the severity of illness of the patient relative to the particular population on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 90 | 90
units on a scale | -0.6 [-0.8 to -0.4] | -0.2 [-0.4 to 0.0]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Placebo; Comparisons between SM-13496 and placebo will be performed by means of a 2-way analysis of covariance (ANCOVA) model with treatment group and study center as factors, and baseline CGI-S score as a covariate. Ninety-five percent (95%) confidence intervals will be constructed using the variability estimates from the ANCOVA model; Test type: Superiority or Other; p < 0.05, ANCOVA

4. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the MADRS (Montgomery Asberg-Depression Scale) Scores
Description: The MADRS is a 10-item rating scale that assesses apparent and reported sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 86 | 83
units on scale | -2.9 [-4.6 to -1.3] | -0.1 [-1.9 to 1.6]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Placebo; Comparisons between SM-13496 and placebo will be performed by means of a 2-way analysis of covariance (ANCOVA) model with treatment group and study center as factors, and baseline MADRS score as a covariate. Ninety-five percent (95%) confidence intervals will be constructed using the variability estimates from the ANCOVA model; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Lurasidone 80 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/90 | 3/90
Other Adverse Events (participants affected / at risk) | 53/90 | 37/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=90) | Placebo (N=90)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Schizophrenia NOS (Psychiatric disorders) | 2 (2) | 1 (1)
Chronic Obstructive Airways Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=90) | Placebo (N=90)
Constipation (Gastrointestinal disorders) | 10 (10) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 15 (15) | 3 (3)
Toothache (Gastrointestinal disorders) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (10) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Akathisia (Nervous system disorders) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 10 (10) | 9 (9)
Sedation (Nervous system disorders) | 9 (9) | 4 (4)
Somnolence (Nervous system disorders) | 10 (10) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No